CLINICAL TRIAL: NCT06832696
Title: Initial Assessment of a Wearable Residual Ultrafiltration Device (RUF-D) to Address Challenges Associated With Inadequate Volume Management in Hemodialysis Patients
Brief Title: Assessment of a Wearable Ultrafiltration Device
Acronym: RUF-D
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Chris McIntyre, Professor of Medicine, Medical Biophysics and Paediatrics,, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15436
Record Dates: First submitted 2025-02-05; First posted 2025-02-18 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Hemodialysis; Ultrafiltration
Keywords: Hemodialysis; Ultrafiltration

STUDY DESIGN:
Intervention Model Description: The proposed study is essentially a feasibility study of both a novel device and therapeutic approach to volume management. Although significant improvement in volume status would be highly impactful, this study will still be deemed a success if initial experience supports that the use of the device is feasible and useable. Efficacy measures relating to the removal of fluid have been chosen to provide objective measures and allow the development of a rational sample size calculation. Investigators aim to study 18 dialysis patients in a prospective unblinded fashion with all recruited participants utilizing the intervention - allowing comparison of primary and secondary end points from baseline assessment and comparison after successful utilization of RUF-D.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients receiving hemodialysis that struggle with fluid removal during dialysis (Experimental): In patients receiving hemodialysis treatment, high amounts of fluid removed in a short time (3-4 hours) can lead to unpleasant symptoms, low blood pressure and can cause bodily stress and organ damage. Leaving this extra fluid in the body also causes undue bodily stress. Investigators need to find gentler, more tolerable ways to remove fluid from patients that need hemodialysis.
  Our investigators have designed and built a new, very small and very simplified device (RUF-D) that can do part of what a dialysis machine does. It doesn't clean the blood or replace the need for dialysis treatments, but it can provide additional and gentle removal of fluid between dialysis treatments which wasn't able to be taken off during a standard treatment session.
  Interventions: Device: RUF-D

INTERVENTIONS:
Device: RUF-D — We have developed a simplified fluid removal device (RUF-D) to address the challenges that patients face with being unable to remove the fluid they need with standard dialysis. Participants 01-09 will receive one week of baseline observation (three HD treatments) with two weeks of supervised intervention using RUF-D post HD on Mondays and Wednesdays for up to six hours (total three-week study).
  Participants 10-18 will receive one week of baseline observation, two weeks of intervention (identical to cohort one above), with an additional week of intervention (total four weeks) where participants will be fitted with the RUF-D (ensuring functionality) before going home with the device in operation for up to six hours twice weekly.

SUMMARY:
Kidney failure is common. In some people the ability of the kidneys to clean poisons out of the blood gets so low they need to be hooked up to a machine three times a week to do it for them. This is called dialysis. Unfortunately, although this treatment removes those waste products, people who need dialysis die much more often than people who don't need dialysis. Dialysis causes extreme stress on the body and leads to many organs being damaged.

Removing fluid from the body quickly causes the equivalent of repeated little heart attacks or little strokes in the brain. Many patients struggle to tolerate having all the fluid that they have drunk since their last dialysis session removed- without unpleasant symptoms of dangerously low blood pressure (which makes the damage worse).

Dialysis treatments can be done more slowly or more often, but that means having to spend a lot more time at the hospital and is difficult for the health system to be able to provide the extra treatment time.

Could extra fluid be removed in between dialysis sessions? Up to now there has not been a way to effectively do this. Investigators have now designed and built an entirely new, very small and very simplified, device that can do part of what a dialysis machine does. It doesn't clean the blood or replace the need for conventional dialysis sessions, but it can provide additional and gentle removal of fluid which wasn't able to be taken off during a standard treatment session.

If this study is successful, it will be the first time that a wearable device has been successfully built and used to take off extra fluid when dialysis patients are not in the hospital. The ability to do this opens up the possibility of, 1) helping to treat patients (both making people feel better and live longer) who can't tolerate getting off all the fluid in the short 3-4 hours they are on the dialysis machine in the hospital, and 2) helping patients who feel OK having the fluid taken off but are silently being subjected to damage to their organs due to the rapid removal, have reduced damage.

DETAILED DESCRIPTION:
The stress of having rapid removal of fluids and waste products condensed into only a 3-4-hour dialysis treatment results in vital organs being repeatedly starved of blood and injured. Our investigators have been at the forefront of demonstrating that the poor outcomes experienced by patients are a direct result from the HD process itself, and these outcomes can be improved by making changes to the dialysis treatment. Our investigators have led the way in showing that taking off too much fluid faster than the body can tolerate causes damage to multiple organ systems; increasing risk of death and symptoms like breathlessness, intense fatigue, long recovery driving cognitive impairment in the brain, and damaging the liver and kidneys (destroying what is left of their own kidney function much faster). Failure to remove the desired amount of fluid during HD is a common occurrence (often due to patient tolerability of treatment time constraints) and is associated with worse QOL, increased HD-induced ischemic injury (heart, brain etc.). Recurrent cardiac injury and loss of contractile function leads to even poorer tolerability of HD and escalating failure to remove accumulated fluid. Patients in this challenging position typically die within 12 months whilst experiencing increased hospitalizations and adversity.

Even a modest difference in how much fluid needs to be removed is of great clinical significance. For instance, reducing the amount that is removed during a four-hour dialysis treatment by only 1 liter reduces the risk of severe heart injury (which effects the overwhelming majority of people) during that treatment.

Our investigators have completed the essential proof-of-concept phase which has allowed refinement of device design and definition of target focus. The principal focus of this next stage was to build a simplified fluid removal system directed at addressing the challenge of patients being unable to remove all the fluid they need to within the standard dialysis treatment.

The proposed study is a feasibility pilot study of both a novel device and therapeutic approach to volume management. Although significant improvement in volume status would be highly impactful, this study will still be deemed a success if initial experience supports that the use of the device is feasible and useable. Investigators intend to study 18 patients in a prospective unblinded fashion, with all recruited patients utilizing the intervention- allowing comparison of primary and secondary end points from baseline assessment and comparison after successful utilization of RUF-D.

ELIGIBILITY:
Inclusion Criteria:

* At least one of the following:

  1. Average per-session IDWG ≥ 4.0% of dry weight in the last month
  2. Inability to consistently achieve dry weight with current HD
  3. Need for additional HD treatments to achieve prescribed dry weight
* HD sessions three times/week
* Age ≥ 18 years
* Dialyzing via central venous access
* Willing and able to provide informed consent

Exclusion Criteria:

* Active infections
* Non-compliance to hemodialysis prescription/schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The device is operational | From enrollment to end of treatment at 4 weeks.
  The device turns on and is able to pump blood through the extracorporeal circuit
The device runs for the desired duration | From enrollment to end of treatment at 4 weeks.
  Achieved by a pre-determined amount of fluid to be removed. If the device runs for the desired length of time to achieve the desired amount of ultrafiltration (eg. 500ml at 2ml/min = 4.2hrs)
The device is comfortable to wear | From enrollment to end of treatment at 4 weeks.
  Comfort will be 'measured' by asking for patient input and feedback

SECONDARY OUTCOMES:
Reduction in Hemodialysis induced acute myocardial injury | From enrolment until the end of treatment at 4 weeks.
  Reduction in number of regional wall motion abnormalities during HD associated with additional interdialytic ultrafiltration, using the RUF-D assessed by echo at each study visit pre and peak dialysis. Regional left ventricular functional assessment will be performed using 2D echocardiography with commercially available equipment (Vivid-I, GE Healthcare) and subsequent automatic analysis of speckle tracked strain curves using automated software (Echo-Pac GE healthcare). Significant stunning will be defined as 50% reduction in regional longitudinal strain.
Reduction in Intradialytic Weight Gain | From enrollment to end of study treatment at 4 weeks.
  Weight measurements to calculate Intradialytic Weight Gain
Reduction in Ultrafiltration Requirements during HD | From enrollment to end of treatment at 4 weeks.
  Weight measurements between treatments

OTHER OUTCOMES:
Change in pre-hemodialysis volume status | From enrollment to end of treatment at 4 weeks.
  Bioimpedance Body Composition Monitor: Bioelectrical impedance analysis (BIA) is based on the principle of detecting resistance to low-level electrical current flows through intracellular and extracellular fluid. Absolute and relative body composition and assessment of total body water (TBW) will be taken using a segmental multifrequency BIA analyzer and Body Composition Monitors (BCM, Fresenius Medical Care, Germany). Measurements will be performed using the standard tetrapolar technique, with electrodes placed unilaterally on wrist and ankle. The analyzer will apply a current, imperceptible to the subject, and software algorithms in the analyzer will measure resistance and reactance and calculate fat-free mass. The extracellular fluid space will be expressed as a proportion of the estimated TBW. The analysis will take place immediately before HD treatments.
Improvement in patient subjective state | From enrollment to end of treatment at 4 weeks.
  A change (from patient's own baseline) in general well-being, pain, sleep, breathing, energy, appetite, itch, restless legs, and recovery time. These parameters will be measured using the LEVIL, an electronic application based visual analog scale.
Changes in hemodynamic response in hemodialysis | From enrollment to end of treatment at 4 weeks.
  The Finometer utilizes a finger-cuff method to detect beat-to-beat changes in digital arterial diameter using an infrared photoplethysmography. The time averaged data is subsequently downloaded to a computer-based analysis program for analysis. The finger-cuff will be placed on the participants middle finger on the non-vascular access arm pre-dialysis and will remain on throughout the entire study visit.
Proportion of treatment successfully delivering intended ultrafiltration volume with RUF-D | From enrollment to end of treatment at 4 weeks.
  Number of treatments that desired ultrafiltration is achieved.
Change in pre-hemodialysis volume status | From enrollment to end of treatment at 4 weeks.
  A vascular ultrasound (IVC diameter) will be completed to check the health of the blood vessels. This involves a test called FMD, which is simple and painless. A cuff is inflated on the arm to temporarily stop blood flow. Once the cuff is released, the ultrasound measures how the artery expands to assess patients' vascular health. The whole process takes about 15 minutes. Minimum IVC diameter can be measured when patient takes a brief sniff or sharp inhale typically, an IVC diameter of >2.0cm and/or with <50% collapsibility upon sharp sniff indicates hypervolemia. IVC ultrasound will be completed at each study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Christopher McIntyre, MBBS DM, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Not yet determined
Supporting Information: Study Protocol
Time Frame: Not yet determined
Access Criteria: Not yet determined